CLINICAL TRIAL: NCT03469427
Title: Reliability of Multislice Computed Tomography Scan in Cases With Facial Nerve Paralysis Due to Temporal Bone Trauma
Brief Title: Multislice Computed Tomography in Cases With Facial Nerve Paralysis Due to Temporal Bone Trauma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sally S Hanna, principle investigator, Assiut University
Other Study IDs: RCTFPTBT
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Facial Nerve Paralysis
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Facial nerve paralysis is a disfiguring complication which occurs in 7-10 % of temporal bone fractures.

The onset of paralysis may be immediate, delayed or undetermined, the latter of which often occurs in unconscious patients with accompanying life-threatening complications.About one fourth has complete paralysis.

DETAILED DESCRIPTION:
Facial nerve paralysis might have variable etiologies apart from idiopathic Bell's palsy, Congenital, infectious, inflammatory, neoplastic, neurological, toxic, iatrogenic and atraumatic causes.

Surgical intervention is indicated if 90-95% loss of function is seen at the very early period on Electroneuronography or if there is axonal degeneration on Electromyography lately with no sign of recovery.

High-resolution multislice computed tomography of the temporal bone is routinely required for evaluation of traumatic facial paralysis. High-resolution multislice computed tomography is known to be the best method for evaluating the intratemporal course of the facial nerve, but it has some limitations as well. Occasionally, the surgeon may encounter facial nerve injuries which have not been revealed in the preoperative computed tomography.

There are limited data in recent medical publications evaluating the diagnostic value of temporal bone High-resolution multislice computed tomography in the evaluation of traumatic facial paralysis. Therefore, in this study,the investigators will compare the findings of preoperative high-resolution multislice computed tomography with surgical findings to determine the diagnostic value of computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* All patients with temporal bone fracture presented with facial nerve paralysis of immediate onset and meet the criteria of facial nerve exploration regardless of age and sex.

Exclusion Criteria:

* Pregnant women.
* Unfit patients for surgery.
* Patients refuse surgical intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of different age groups presented with facial nerve paralysis due to temporal bone trauma
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Patients who suffer from facial nerve paralysis due to temporal bone trauma will be diagnosed by using multislice computed tomography | up to 2 years
  Evaluation the reliability of multislice computed tomography in the assessment of facial nerve paralysis due to temporal bone trauma

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided